CLINICAL TRIAL: NCT03752879
Title: The Association Between Fundal Pressure in Second Stage of Labor (Kristeller Maneuver) and and Pelvic Floor Trauma After Vaginal Delivery
Brief Title: The Association Between Kristeller Maneuver and Pelvic Floor Trauma After Vaginal Delivery
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BezmialemVU Fundal Pressure
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Labor Complication; Avulsion
Keywords: Kristeller maneuver,LAM avulsion,3D transperineal ultrasoun
MeSH Terms: conditions — Obstetric Labor Complications; Fractures, Avulsion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case (Kristaller Group): Group of kristeller maneuver applied in the second stage of labor due to clinical necessity.
  Interventions: Procedure: Fundal Pressure
- Control (no Kristaller Group): The control group not required to kristeller maneuver

INTERVENTIONS:
Procedure: Fundal Pressure — Fundal Pressure to assist the vaginal delivery to shorten the second stage of labor
  Groups: Case (Kristaller Group)

SUMMARY:
We want to investigate the association between fundal pressure in the second stage and the risk of levator ani muscle (LAM) injury.

DETAILED DESCRIPTION:
We will recruit women immediately following their first vaginal delivery. Women who underwent Kristeller maneuver will be recruit as cases. For each case, a control (no fundal pressure) will be recruit matched by BMI, second stage duration and birthweight. All women will be invited to undergo a postpartum 3D transperineal ultrasound (TPUS). The main outcome measure will be the presence of LAM avulsion at 3D TPUS. TPUS results will be compared between cases and controls.

ELIGIBILITY:
Inclusion Criteria:

* First delivery
* Term pregnancy (37-41w)

Exclusion Criteria:

* Instrumental vaginal delivery
* Multifetal pregnancy
* Previous vaginal or cesarean delivery
* Refused consent and uncooperative patient for effective Valsalva maneuver
* Handicap in lithotomy position
* Women without regular and active contractions
* Epidural analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — biological female gender
Study Population: Over 18 years old ,term primiparous women with singleton pregnancies and vaginal delivery.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-05-18 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
levator ani muscle (LAM) injury | 24 hour
  The aim of the study is to investigate levator ani muscle (LAM) injury, loss of tenting, biometric measurements of LAM and genital hiatus after vaginal delivery and investigate the association between fundal pressure in the second stage of labor (Kristeller maneuver).
  All recruited women will be invited to undergo a transperineal 3D ultrasound (TPUS) scan at 24 hours after delivery. we will acquire two 3D volumes for each patient: one under maximum pelvic floor muscle contraction (PFMC) and the other under maximum Valsalva's maneuver. Ballooning" will diagnosed with a pelvic hiatal area of more than 25 cm2 during maximum Valsalva. A complete avulsion of the puborectalis muscle will diagnose if an abnormal insertion of the muscle will be detected on all three central slices. We will use a levator-urethral gap more than 2.5 cm to define an abnormal insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takmaz T, Aydin S, Gorchiyeva I, Karasu AFG. The usual suspect: cross-sectional study of fundal pressure at second stage of delivery and the association with pelvic floor damage. Int Urogynecol J. 2021 Jul;32(7):1917-1924. doi: 10.1007/s00192-020-04523-x. Epub 2020 Sep 9. PMID 32902763